CLINICAL TRIAL: NCT05023304
Title: In Clinic Optometrist Insertion of Dextenza Prior to Cataract Surgery
Acronym: Prepare
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vance Thompson Vision (Other)
Collaborators: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: The Prepare Study
Record Dates: First submitted 2021-08-02; First posted 2021-08-26 (Actual); Results first posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Calcium Dobesilate; prednisolone acetate

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A Dextenza (Experimental): Randomized to dexamethasone ophthalmic insert 0.4mg placed prior to cataract surgery, on the day of surgery.
  Interventions: Drug: Dextenza 0.4Mg Ophthalmic Insert
- Group B Topical Prednisolone (Active Comparator): Randomized to topical prednisolone acetate 1% four times per day for one week, three times per day for one week, two times per day for one week, and one time per day for one week starting after 4 hours after surgery.
  Interventions: Drug: Topical prednisolone acetate

INTERVENTIONS:
Drug: Dextenza 0.4Mg Ophthalmic Insert — The insert, containing 0.4 mg of active pharmaceutical product, is placed within the canaliculus to provide a sustained and tapered delivery of drug to the ocular surface over 30 days after a one-time insertion. The attributes of the insert reduce the risks for improper corticosteroid tapering and unwanted peaks and troughs in drug concentration.
  Arms: Group A Dextenza
Drug: Topical prednisolone acetate — Standard of care topical drop regimen with four week taper
  Arms: Group B Topical Prednisolone

SUMMARY:
To evaluate the clinical outcomes with optometrist pre-surgical insertion of DEXTENZA in the clinical office setting in patients undergoing same-day cataract surgery compared to standard of care steroid therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older, undergoing routine, uncomplicated, sequential bilateral cataract surgery.
* Willing and able to comply with clinic visits and study related procedures
* Willing and able to sign the informed consent form

Exclusion Criteria:

* Patients under the age of 18.
* Patients who are pregnant (must be ruled out in women of childbearing age with pregnancy test).
* Active infectious ocular or systemic disease.
* Patients with active infectious ocular or extraocular disease.
* Patients actively treated with local or systemic immunosuppression including systemic corticosteroids.
* Patients with known hypersensitivity to Dexamethasone.
* Patients with severe disease that warrants critical attention, deemed unsafe for the study by the investigator.
* Patients with proliferative diabetic retinopathy or uncontrolled diabetes as deemed by an A1C > 10.0.
* Patients with a history of ocular inflammation or macular edema.
* Patients with a pre-existing epiretinal membrane (ERM)
* Patients with allergy or inability to receive intracameral antibiotic.
* Patients on systemic non-steroidal anti-inflammatory drugs (NSAID) greater than 1,200 mg/day The PREPARE Study (V1) February, 2021 Page 27 CONFIDENTIAL
* Patients with a corticosteroid implant (i.e. Ozurdex).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitch Ibach, OD, Principal Investigator — Vance Thompson Vision
Locations (1):
- Vance Thompson Vision, Sioux Falls, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Contralateral eye study with randomization of one eye receiving a dexamethasone ophthalmic insert 0.4mg and the other eye receiving topical prednisolone acetate 1% four times daily for one week, three times daily for one week, two times daily for one eye, and then one time daily for one week.
Pre-assignment Details: 60 eyes of 30 patients enrolled
Units Other Than Participants: Eyes
Groups:
- Group A Dextenza Ophthalmic Insert 0.4mg: Randomized to dexamethasone ophthalmic insert 0.4mg placed prior to cataract surgery, on the day of surgery.
  Dextenza 0.4Mg Ophthalmic Insert: The insert, containing 0.4 mg of active pharmaceutical product, is placed within the canaliculus to provide a sustained and tapered delivery of drug to the ocular surface over 30 days after a one-time insertion. The attributes of the insert reduce the risks for improper corticosteroid tapering and unwanted peaks and troughs in drug concentration.
- Group B Topical Prednisolone Acetate 1%: Randomized to topical prednisolone acetate 1% four times per day for one week, three times per day for one week, two times per day for one week, and one time per day for one week starting after 4 hours after surgery.
  Topical prednisolone acetate: Standard of care topical drop regimen with four week taper
Period: Overall Study
Arm/Group | Group A Dextenza Ophthalmic Insert 0.4mg | Group B Topical Prednisolone Acetate 1%
Started | 30; 30 Eyes | 30; 30 Eyes
Completed | 30; 30 Eyes | 30; 30 Eyes
Not Completed | 0; 0 Eyes | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Population: Contralateral eye study with randomization where one eye received a dexamethasone ophthalmic insert 0.4mg and the other received topical prednisolone acetate 1% four times daily for one week, three times daily for one week, then two times daily for one week, and then one time daily for one week
Units Other Than Participants: Eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A Dextenza | Group B Topical Prednisolone | Total
Number analyzed (Participants) | 30 | 30 | 60
Number analyzed (Eyes) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (0.389) | 67 (0.389) | 67 (0.389)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 34
  Male | 13 | 13 | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Pain Score 0-10 [Mean (Full Range); unit: units on a scale] — second measure in the primary outcome was mean pain score as measured by Visual Analog Score numerical grading scale 0-10 at post-op day 1, day 7, and week 4.
  units on a scale | 2 [0 to 10] | 2 [0 to 10] | 2 [0 to 10]

OUTCOME MEASURES:

1. Primary Outcome: Mean Anterior Chamber Cell/Flare Score
Description: Mean anterior chamber cell/flare score measured by Slit Lamp Biomicroscopy evaluation using grading scale of 0 to 4 +. The scale used is called the (Standardization of Uveitis Nomenclature) SUN Working Group Grading Scheme. AC cell grading schema. The SUN Working Group defined their two AC grading schemas around these two findings. Importantly, for all grading schemas discussed in this article, an improvement in inflammation is a two-step decrease in grade. A worsening of inflammation occurs with a two-step increase in grade. Grade 0 = 0 cells per high power field or HPF; Grade 0.5+ = 1-5 cells HPF; 1+ = 6-15 HPF; 2+ = 16-25 HPF; 3+ = 26-50 HPF; 4+ >50.
Time Frame: Post-op Day 1
Population: Contralateral eye study of 30 patients. A total of 60 eyes analyzed with 30 eyes randomized to each group.
Measure: Mean (Full Range); unit: Units on a scale
Units Other Than Participants: eyes
Arm/Group | Group A Dextenza | Group B Topical Prednisolone
Number analyzed (Participants) | 30 | 30
Number analyzed (eyes) | 30 | 30
Units on a scale | 1.06 [0 to 4] | 1.15 [0 to 4]

2. Primary Outcome: Mean Anterior Chamber Cell/Flare Score
Description: Mean anterior chamber cell/flare score measured by Slit Lamp Biomicroscopy evaluation using grading scale of 0 to 4 +. The scale used is called the (Standardization of Uveitis Nomenclature) SUN Working Group Grading Scheme. AC cell grading schema. The SUN Working Group defined their two AC grading schemas around these two findings. Importantly, for all grading schemas discussed in this article, an improvement in inflammation is a two-step decrease in grade. A worsening of inflammation occurs with a two-step increase in grade. Grade 0 = 0 cells per high power field or HPF; Grade 0.5+ = 1-5 cells HPF; 1+ = 6-15 HPF; 2+ = 16-25 HPF; 3+ = 26-50 HPF; 4+ >50. The higher the HPF, the more inflammation that can negatively impact a patient's outcome.
Time Frame: Post-op Day 7
Population: Contralateral eye study of 30 patients. A total of 60 eyes analyzed with 30 eyes randomized to each group.
Measure: Mean (Full Range); unit: score on a scale
Units Other Than Participants: eyes
Arm/Group | Group A Dextenza | Group B Topical Prednisolone
Number analyzed (Participants) | 30 | 30
Number analyzed (eyes) | 30 | 30
score on a scale | 0.25 [0 to 4] | 0.22 [0 to 4]

3. Primary Outcome: Number of Eyes With No Cell or Flare Measured
Description: as for outcome 2
Time Frame: post-op Week 4.
Population: Contralateral eye study of 30 patients. A total of 60 eyes analyzed with 30 eyes randomized to each group.
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Group A Dextenza | Group B Topical Prednisolone
Number analyzed (Participants) | 30 | 30
Number analyzed (eyes) | 30 | 30
eyes | 30 | 28

4. Primary Outcome: Mean Pain Score
Description: Mean pain score measured by Visual Analog Score numerical grading scale 0(minimum)-10(maximum) 0= absence of pain 10 = highest possible pain A higher number indicates a higher pain value which may impact a subject's outcomes.
Time Frame: Post-op Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group A Dextenza | Group B Topical Prednisolone
Number analyzed (Participants) | 30 | 30
Participants
  Pain score 0 | 23 | 23
  Pain score 1 | 2 | 2
  Pain score 2 | 2 | 3
  Pain score 3 | 2 | 2
  Pain score 4 | 1 | 0

5. Primary Outcome: Patient Tolerability (Defined as Patient Preference)
Description: As measured by adapted COMTOL (Comparison of Ophthalmic Medications for Tolerability) Questionnaire. The COMTOL questionnaire is designed to assess the tolerability of topical ophthalmic medications. It consists of several elements that help evaluate the frequency, severity, and impact of common side effects: Section 1: Ocular Side Effects; Section 2: Local Side Effects; Section 3: Visual Function; Section 4: Impact on Quality of Life. Likert scale is used to measure each question. 1=Never, 2=Rarely, 3=Sometimes, 4 = Often, 5= Always. A higher score suggests that the medication is less well-tolerated and may be negatively impacting the patient's daily activities and overall well-being.
Time Frame: Post-op Week 4
Population: 30 patients in each cohort or 60 eyes
Measure: Count of Participants; unit: Participants
Groups:
- All Study Participants: All Study Participants who completed the questionnaire
Arm/Group | All Study Participants
Number analyzed (Participants) | 30
Participants
  Preferred Dexamethasone Inserts | 29
  Preferred Preferred topical prednisolone acetate | 0
  No Preference | 1

6. Secondary Outcome: Number of Participants With Increased Intraocular Pressure (IOP) >10mmHg Above Baseline
Description: Intraocular pressure as measured by Goldmann Applanation Tonometer; Total number of Participants with Increased IOP >10mmHg above baseline. Normal intraocular pressure (IOP) is generally considered to be between 10 and 21 millimeters of mercury (mmHg). However, it's important to note that this is just a general range, and individual values can vary. A higher IOP may negatively impact a subject's outcome.
Time Frame: postop Day 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group A Dextenza | Group B Topical Prednisolone
Number analyzed (Participants) | 30 | 30
Participants | 1 | 0

7. Secondary Outcome: Number of Participants With Increased Intraocular Pressure (IOP) >10mmHg Above Baseline
Description: as for outcome 6
Time Frame: Postop Day 7
Measure: Count of Participants; unit: Participants
Arm/Group | Group A Dextenza | Group B Topical Prednisolone
Number analyzed (Participants) | 30 | 30
Participants | 0 | 0

8. Secondary Outcome: Number of Participants With Increased Intraocular Pressure (IOP) >10mmHg Above Baseline
Description: Intraocular Pressure as measured by Goldmann Applanation Tonometer, Total number of Participants with increased IOP > 10mmHg above baseline. Normal intraocular pressure (IOP) is generally considered to be between 10 and 21 millimeters of mercury (mmHg). However, it's important to note that this is just a general range, and individual values can vary. A higher IOP may negatively impact a subject's outcome.
Time Frame: postop Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Group A Dextenza | Group B Topical Prednisolone
Number analyzed (Participants) | 30 | 30
Participants | 0 | 0

9. Secondary Outcome: Number of Participants With Post-operative Cystoid Macular Edema (CME)
Description: Cystoid Macular Edema (CME) as measured by optical coherence tomography (OCT); Total number of study participants with post-operative CME.
Time Frame: post-op Week 4
Measure: Count of Participants; unit: Participants
Arm/Group | Group A Dextenza | Group B Topical Prednisolone
Number analyzed (Participants) | 30 | 30
Participants | 0 | 0

10. Secondary Outcome: Physician Ease of Use
Description: Physician Ease of Use Survey following dexamethasone intracanalicular placement on Surgical Visit on Scale of 0-10 with 10 being most complex (0= minimum value or not complex and 10= maximum complexity). A higher number indicates a worse outcome.
Time Frame: Day 0
Population: Not applicable to Group B
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | Group A Dextenza | Group B Topical Prednisolone
Number analyzed (Participants) | 30 | 0
Score on a scale | 3.9 [0 to 10] |

11. Secondary Outcome: Eye Drop Burden Reported by Participants
Description: Eye Drop Burden Questionnaire numerical grading scale 8 questions on scale of 1-5 totaling a maximum score of 40.
  Likert scale used: 1 Very easy, 2. Easy 3. Neither easy nor difficult 4. Difficult 5. Very difficult Low Burden=8-18 Moderate Burden=19-29 High Burden= 30-40 A higher number score indicates a negative outcome for a subject.
Time Frame: Post-op Day 7
Population: 1 patient did not complete questionnaire. Patients were not asked to differentiate between eyes when answering the eye drop burden questionnaire
Measure: Count of Participants; unit: Participants
Groups:
- 30 Participants: Both the Dexamethasone insert group and topical prednisone group remained on standard of care antibacterial and nonsteroidal anti-inflammatory topical drops. Patients were instructed to use moxifloxacin four times daily for two weeks and topical nonsteroidal anti-inflammatory for one month. Patients were not asked to differentiate between eyes when answering the eye drop burden questionnaire
Arm/Group | 30 Participants
Number analyzed (Participants) | 29
Participants
  Low burden (maximum score between 8-18) | 27
  Moderate burden (maximum score between 19-29) | 2
  High burden (maximum score between 30-40) | 0

12. Secondary Outcome: Eye Drop Burden Reported by Participants
Description: Eye Drop Burden Questionnaire numerical grading scale 8 questions on scale of 1-5 totaling a maximum score of 40.
  Likert scale used: 1 Very easy, 2. Easy 3. Neither easy nor difficult 4. Difficult 5. Very difficult Low Burden=8-18 Moderate Burden=19-29 High Burden= 30-40 A higher score is considered a worse outcome for a subject.
Time Frame: post-op Week 4. Patients were not asked to differentiate between eyes when answering the eye drop burden questionnaire
Measure: Count of Participants; unit: Participants
Groups:
- 30 Participants: Each group remained on standard of care antibacterial and nonsteroidal anti-inflammatory topical drops. Patients were instructed to use moxifloxacin four times daily for two weeks and topical nonsteroidal anti-inflammatory for one month. Patients were not asked to differentiate between eyes when answering the eye drop burden questionnaire
Arm/Group | 30 Participants
Number analyzed (Participants) | 30
Participants
  Low burden (maximum score between 8-18) | 28
  Moderate burden (maximum score between 19-29) | 2
  High burden (maximum score between 30-40) | 0

ADVERSE EVENTS:
Time Frame: Data was collected out to 3 months post-operative
Arm/Group | Group A Dextenza | Group B Topical Prednisolone
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/04/NCT05023304/Prot_001.pdf
  • Informed Consent Form (2021-08-03): https://cdn.clinicaltrials.gov/large-docs/04/NCT05023304/ICF_002.pdf